CLINICAL TRIAL: NCT02064881
Title: Effect of Metformin Glycinate on Postprandial Lipemia, Glycemic Control and Oxidation Markers in Type 2 Diabetes Patients
Brief Title: Efficacy Study of Metformin Glycinate on Postprandial Lipemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMMET_LP001
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes
Keywords: Postprandial lipemia; Diabetes; Metformin glycinate; oxidized LDL
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin glycinate (Experimental): 620mg tablets of metformin glycinate: 1 tablet by mouth at night for 3 days, 1 tablet in the morning and evening for 3 days, 1 tablet in the morning and 2 tablets in the evening for 3 days and 2 tablets in the evening and 2 tablets in the morning until the end of the study.
  Total study dose: 1240mg every 12 hours.
  Interventions: Drug: Metformin glycinate
- metformin hydrochloride (Active Comparator): 500mg tablets of metformin hydrochloride:1 tablet by mouth at night for 3 days, 1 tablet in the morning and evening for 3 days, 1 tablet in the morning and 2 tablets in the evening for 3 days and 2 tablets in the evening and 2 tablets in the morning until the end of the study.
  Total study dose: 1000mg every 12 hours.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin glycinate — All patients are going to begin the treatment with one tablet orally at night, 30 minutes before dinner (1 tablet of 620 mg glycinate metformin or one 500 mg tablet of metformin hydrochloride) and the dose will be administrated every 3 days to complete the dose of 2 tablets in the morning 30 minutes before breakfast and 2 tablets in the evening 30 minutes before dinner (1240 mg metformin glycinate every 12 hours or 1000 mg metformin hydrochloride every 12 hrs) .
  Other Names: DMMET-01
  Arms: metformin glycinate
Drug: Metformin Hydrochloride — All patients are going to begin the treatment with one tablet orally at night, 30 minutes before dinner (1 tablet of 620 mg glycinate metformin or one 500 mg tablet of metformin hydrochloride) and the dose will be administrated every 3 days to complete the dose of 2 tablets in the morning 30 minutes before breakfast and 2 tablets in the evening 30 minutes before dinner (1240 mg metformin glycinate every 12 hours or 1000 mg metformin hydrochloride every 12 hrs)
  Other Names: HCL MET
  Arms: metformin hydrochloride

SUMMARY:
The aim of this study is to evaluate the effect of metformin glycinate vs metformin hydrochloride on postprandial lipemia. 72 patients will be included, they will be randomized and assigned into one of the two treatment groups: metformin glycinate 1240 mg BID or metformin hydrochloride 1000 mg BID (36 patients per group). The patients will be followed for 4 months.

Blood count, blood chemistry, liver profile, lipid profile, HbA1c, apolipoprotein B, oxidized LDL, fibroblast growth factor 21, leptin, adiponectin, C-reactive protein, free fatty acids, fibrinogen, Goodpasture Binding Protein (GPBP) and antioxidant activity of plasma will be measured at baseline and 4 months.

Additionally, after a structured meal, the following parameters will be measured: glucose, insulin, triglycerides, apolipoprotein B and oxidized LDL. (baseline and 4 months). Throughout the study adverse events will be documented.

DETAILED DESCRIPTION:
Main objective: To compare the effect of metformin glycinate with metformin hydrochloride postprandial lipemia (area under the curve of triglycerides)

Study group

Tablets of 620 mg of metformin glycinate. Scaling: 1 tablet at night for 3 days, followed by 1 tablet in the morning and 1 tablet at night for 3 days, followed by 1 tablet in the morning and 2 tablets in the evening for 3 days and finally, 2 tablets in the morning and 2 tablets in the evening to complete the study. Final study dose 1240 mg every 12 hours.

Comparative group

500 mg tablets of metformin hydrochloride. Scaling: 1 tablet at night for 3 days, followed by 1 tablet in the morning and 1 tablet at night for 3 days, followed by 1 tablet in the morning and 2 tablets in the evening for 3 days and finally, 2 tablets in the morning and 2 tablets in the evening to complete the study. Final study dose 1000 mg every 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Between 35 and 65 years old
* Patients with type 2 diabetes within two years of diagnosis according to the ADA criteria
* Overweight patients (BMI between 25.5 and 29.9 kg/m2) or with grade 1 obesity (BMI between 30.0 and 34.9 kg/m2), according to WHO classification
* Low HDL levels: <50 in women and <40 mg/dL in men
* Hypertriglyceridemia: >150 and less than 300 mg/dL
* Patients who had not taken antidiabetes drug treatment or with diet and exercise treatment, or with metformin or DPP4 inhibitor monotherapy
* HbA1c between 6.5 and 8.5%.
* Creatinine clearance >60 ml/min (calculated by Cockcroft and Gault)
* Informed consent form signed.
* Women using contraception.

Exclusion Criteria:

* Patients with other types of diabetes (type 1, LADA, MODY, etc.).
* Patients with primary dyslipidemia.
* Patients with poorly substituted hypothyroidism TSH > 5 mU/mL.
* Patients hospitalized in the last month.
* Patients with a disease of poor short-term prognosis
* Patients with autoimmune or rheumatic diseases.
* Patients with acute infection or febrile illness.
* History of chronic liver disease or ALT or AST ≥ 2.0 times the upper limit of normal, or GGT ≥ 3 times the upper limit of normal.
* Patients with any other chronic disease, for example: HIV, rheumatic diseases.
* Pregnant or positive pregnancy test.
* Women who are breastfeeding.
* Patients in another research project.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in postprandial lipemia at 4 months | baseline, 4 months

SECONDARY OUTCOMES:
Change in oxidized LDL at 4 months | baseline, 4 months
Change in FGF-21 levels at 4 months | baseline, 4 months
Change in A1C at 4 months | baseline, 4 months
Change in alanine aminotransferase at 4 months | baseline, 4 months
Change in uric acid at 4 months | baseline, 4 months
Number of Participants with Serious and Non-Serious Adverse Events | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Gómez, Doctor, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas Y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Schramm TK, Gislason GH, Vaag A, Rasmussen JN, Folke F, Hansen ML, Fosbol EL, Kober L, Norgaard ML, Madsen M, Hansen PR, Torp-Pedersen C. Mortality and cardiovascular risk associated with different insulin secretagogues compared with metformin in type 2 diabetes, with or without a previous myocardial infarction: a nationwide study. Eur Heart J. 2011 Aug;32(15):1900-8. doi: 10.1093/eurheartj/ehr077. Epub 2011 Apr 6. PMID 21471135
- [Background] Masoudi FA, Inzucchi SE, Wang Y, Havranek EP, Foody JM, Krumholz HM. Thiazolidinediones, metformin, and outcomes in older patients with diabetes and heart failure: an observational study. Circulation. 2005 Feb 8;111(5):583-90. doi: 10.1161/01.CIR.0000154542.13412.B1. PMID 15699279
- [Background] Roussel R, Travert F, Pasquet B, Wilson PW, Smith SC Jr, Goto S, Ravaud P, Marre M, Porath A, Bhatt DL, Steg PG; Reduction of Atherothrombosis for Continued Health (REACH) Registry Investigators. Metformin use and mortality among patients with diabetes and atherothrombosis. Arch Intern Med. 2010 Nov 22;170(21):1892-9. doi: 10.1001/archinternmed.2010.409. PMID 21098347